CLINICAL TRIAL: NCT06660251
Title: Trimethylamine-N-oxide After Animal Food - Effects of Gut Microbiota in Subjects with and Without Metabolic Syndrome
Brief Title: Effect of Meat and Egg on TMAO in Plasma and Urine in Subjects with and Metabolic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Mohammed Hefni, Assoc Prof, Linnaeus University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-04354
Record Dates: First submitted 2024-10-07; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic syndrome; TMAO; Gut microbiota; Egg and meat; Plasma; Urine
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized, crossover intervention with two active groups (subjects with and without MetS) using two test foods (egg and meat, with high content of TMAO precursors) was carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects with MetS (Active Comparator): Subjects with a minimum of three criteria according to NCEP-ATP III. Subjects were administered in randomized order after overnight fasting a test food. Test days were on two separate occasions around 2 weeks apart.
  Egg intervention: three hard-boiled eggs. Meatball intervention: 170 g meatballs.
  Interventions: Other: Egg intervention; Other: Meatball intervention
- Subjects without MetS (Active Comparator): Subjects, apparently healthy, with normal BMI, blood pressure, waist circumference (see inclusion criteria). Subjects were administered in randomized order after overnight fasting a test food. Test days were on two separate occasions around 2 weeks apart.
  Egg intervention: three hard-boiled eggs. Meatball intervention: 170 g meatballs.
  Interventions: Other: Egg intervention; Other: Meatball intervention

INTERVENTIONS:
Other: Egg intervention — Oral administration of three hard-boiled eggs to be ingested within 15 minutes on one occasion.
Other: Meatball intervention — Oral intervention with 170 g meatballs to be ingested within 15 minutes on one occasion.

SUMMARY:
The purpose of this clinical trial is to investigate in subjects with and without metabolic syndrome how meals of choline- and carnitine-rich foods (eggs and meat) affect the trimethylamine-N-oxide (TMAO) concentration in blood and urine in relation to the gut microbiota composition.

In response to the subjects´ gut microbiota, the concentrations of TMAO in the plasma and urine of subjects with and without metabolic syndrome (MetS) after ingesting choline- and carnitine-rich foods will be compared.

On two occasions, participants will receive after overnight fasting meatballs (170 g) or three hard-boiled eggs. Blood will be collected before ingestion and over 6 hours after test food consumption.

DETAILED DESCRIPTION:
There is a growing interest in the role of the intestinal microbiota in the global metabolism of their host. Trimethylamine-N-oxide (TMAO), a metabolite linked to the gut microbiota, has recently emerged as a risk metabolite for cardiovascular disease.

The gut microbiota composition was reported to be altered in MetS. After ingestion of foods high in trimethylamine moieties, postprandial TMAO in blood may differ between subjects with and without MetS because of their different microbiota profiles.

Aim of the study is to investigate in subjects with and without MetS the postprandial TMAO concentrations in blood and urine in association with the gut microbiota profile after ingestion of choline- and L-carnitine-rich foods.

Thirty-three subjects aged 18-75 years with (n=12) or without MetS (n=21) were recruited.

Subjects received on two occasions, after overnight fasting, either three hard-boiled eggs or 170 g meatballs.

Blood samples were collected (before ingestion of food, and at 30, 60, 120, 240, and 360 minutes after ingestion). A composite urine sample was collected over 6 hours. A feces sample was collected on the day before the first intervention.

Concentrations of TMAO, trimethylamine, betaine, choline, L-carnitine, acetyl-L-carnitine, and creatinine were measured UPLC-MRM-MS. The incremental area under the curve (iAUC) was calculated for each compound.

TMAO, trimethylamine, betaine, choline, L-carnitine, acetyl-L-carnitine, and creatinine were analyzed in composite urine samples using UPLC-MRM-MS.

Gut microbiome analysis was done by full 16S rRNA gene sequencing using the Oxford Nanopore Technology.

ELIGIBILITY:
Inclusion criteria for all subjects with and without MetS:

* Age = 18-75y
* Plasma creatinine value within the age-related reference range
* No history of acute or chronic diseases (e.g. diabetes or bowel disease)
* No use of vitamin or mineral supplements, no medication with antibiotics 2 months before recruitment and during the study
* Non-smoker
* Not consuming a special diet (vegetarian)
* No pregnancy, planned conception, or lactation
* No participation in another study.

Inclusion criteria for subjects without MetS:

* Normal BMI (18.6 to 29.0 kg / m 2 )
* Blood counts within reference ranges
* Normal ranges for liver enzymes (P-ALAT, P-AST, P-ALP), blood status, plasma triglycerides, plasma HDL cholesterol, plasma cholesterol, plasma glucose

Inclusion criteria for subjects with MetS:

A minimum of three of the following criteria according the National Cholesterol Education Program Adult Treatment Panel (NCEP-ATP III):

* Waist size > 102 cm in men, > 88 cm in women
* Fasting plasma glucose ≥ 5.6 mmol /l
* Triglycerides > 1.7 mmol / l or treatment
* HDL 1.03 mmol / l in men, 1.29 mmol / l in women or treatment
* Blood pressure ≥ 130 / 85 mm Hg or medication. A value of B-HbA1c in the age-related reference range will be used to exclude diabetes.

Exclusion criteria for all research subjects :

* Smoker
* Pregnancy, planned conception, or lactation
* Medical treatment with antibiotics 2 months before recruitment and during the study
* Use of dietary supplements 2 weeks before and during the study
* Use of probiotics 2 months before and during the study
* Following a special diet (eg vegan, vegetarian, weight loss)
* Participation in another study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
TMAO and related metabolite concentrations (micromole per litre) in plasma | Metabolite concentrations in plasma samples collected before ingestion of test food and after ingestion at 30, 60, 120, 240, and 360 minutes are used for calculation the incremental area under the curve.
  TMAO and related metabolites (trimethylamine, betaine, choline, L-carnitine, and acetyl-L-carnitine) were analyzed by UPLC-MRM-MS in plasma samples collected before ingestion of test food and after ingestion at 30, 60, 120, 240, and 360 minutes.
TMAO and related metabolite concentrations (micromole per litre) in urine | Post-dose sample over a 6-hours period.
  TMAO and related metabolites (trimethylamine, betaine, choline, L-carnitine, and acetyl-L-carnitine) were analyzed by UPLC-MRM-MS in a composite urine sample collected during 6 hours post-dose.

SECONDARY OUTCOMES:
Gut microbiota composition | The day before the first intervention day.
  Gut microbiota composition in a stool sample collected on the day before the first intervention was analyzed by a full 16S rRNA gene sequencing kit from Oxford Nanopore Technology.
Blood glucose and glycated hemoglobin | At screening (before intervention).
  Fasting blood glucose and glycated hemoglobin (millimoles per liter mmol/l) were analyzed at screening.
Plasma lipid profile | At screening (before intervention).
  Plasma cholesterol, plasma high-density lipoprotein cholesterol, plasma cholesterol, and plasma triglycerides concentrations (millimoles per liter mmol/l) were analyzed at screening.
Body mass index (BMI) | At screening (before intervention).
  Weight in kilograms and height in meters were measured at screening and used to calculate BMI in kilograms per square.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Hefni, Assoc Prof, Principal Investigator — Linnaeus University
Locations (1):
- Faculty of Health and Life Sciences, Linnaeus University, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data as all data will be presented in the main article through tables and figures or in the supplementary material as mean ± standard deviation. However, individual data will be made available upon reasonable request.